CLINICAL TRIAL: NCT02486133
Title: A Prosp., Multic., Randomized, Open-label Trial to Assess the Safety, Tolerability and Efficacy of Dual Therapy With Boosted Darunavir + Dolutegravir When Switching From SOC ART in HIV-patients With Sustained Virological Suppr.
Brief Title: Dual Therapy With Boosted Darunavir + Dolutegravir
Acronym: Dualis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUA-1463-SPI-0320-I
Record Dates: First submitted 2015-06-15; First posted 2015-07-01 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2019-04

CONDITIONS: HIV-Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir; dolutegravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; abacavir, lamivudine drug combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: boosted darunavir (bDRV) plus dolutegravir (DTG; 2DR) (Experimental): Prezista & Norvir & Tivicay
  Interventions: Drug: Prezista; Drug: Norvir; Drug: Tivicay
- B: bDRV plus 2 nucleoside reverse-transcriptase inhibitors (NRTIs; 3DR) (Active Comparator): Prezista & Norvir & Truvada or Prezista & Norvir & Kivexa or Prezista & Norvir & Descovy
  Interventions: Drug: Prezista; Drug: Norvir; Drug: Truvada; Drug: Kivexa; Drug: Descovy

INTERVENTIONS:
Drug: Prezista — once daily
  Other Names: Darunavir
Drug: Norvir — once daily
  Other Names: Ritonavir
Drug: Tivicay — once daily
  Other Names: Dolutegravir
  Arms: A: boosted darunavir (bDRV) plus dolutegravir (DTG; 2DR)
Drug: Truvada — once daily
  Other Names: Tenofovir disaproxil fumarat/emtricitabine
  Arms: B: bDRV plus 2 nucleoside reverse-transcriptase inhibitors (NRTIs; 3DR)
Drug: Kivexa — once daily
  Other Names: Abacavir/Lamivudine
  Arms: B: bDRV plus 2 nucleoside reverse-transcriptase inhibitors (NRTIs; 3DR)
Drug: Descovy — once daily
  Other Names: Tenofovir alafenamid / emtricitabine
  Arms: B: bDRV plus 2 nucleoside reverse-transcriptase inhibitors (NRTIs; 3DR)

SUMMARY:
A switch strategy to investigate whether a dual therapy with Ritonavir-boosted (RTV) Darunavir (DRV) + Dolutegravir (DTG) over 48 weeks is non-inferior to a continuous standard of care therapy with RTV-boosted DRV in combination with 2 Nucleosidic Reverse Transcriptase Inhibitors (NRTIs) in HIV patients, who are on a stable antiretroviral therapy (ART) with RTV-boosted DRV in combination with 2 NRTIs.

DETAILED DESCRIPTION:
Modern combination antiretroviral therapy (cART) leads to well-controlled HIV infection with a potentially normal life expectancy. Nucleosidic reverse transcriptase inhibitors (NRTIs) play a major role as "ART backbone" and are essential antiretroviral agents according to current European and WHO HIV treatment guidelines. However, NRTI use can be associated with substantial side effects, e.g. bone and kidney toxicity, lipotoxicity and mitochondrial toxicity and can put patients at serious risk. Especially long-term NRTI-exposure is a risk factor for these often cumulative side effects, since the standard of care (SOC) therapy with the different NRTIs consists of the combination of multiple substances. Furthermore NRTI resistances may emerge over time and limit treatment options for pre-treated HIV patients.

As a consequence, alternative NRTI free (so called "nuke sparing") therapy options have been evaluated in different studies but were associated with less virologic therapeutic success and higher rates of therapy induced resistance compared to standard regimens in ART naïve patients. This is particularly true for patients with a high baseline viral load.

As an alternative to NRTI-based therapy options, Ritonavir-boosted protease inhibitor (PI/r)-based nuke-sparing dual therapies have been studied widely, mostly in combination with the integrase inhibitor (INI) Raltegravir (RAL). In this setting, the PI was not fully capable to prevent the development of INI resistant viruses.

The HIV protease inhibitor Darunavir (DRV) and the novel INI Dolutegravir (DTG) are both very potent anchor drugs with a high barrier to resistance. Due to a favourable side-effect profile, a once-daily (QD) formulation and its virological potency, DRV is currently one of the most frequently used PIs in Europe and the USA. In addition, the new, once-daily administrable integrase inhibitor DTG showed an excellent tolerability profile as well as a high resistance barrier.

The nuke-free combination of DTG (50 mg) with the Ritonavir (/r)- or Cobicistat-boosted protease inhibitor DRV (800 mg) may offer a favorable safety and efficacy profile with the advantage of QD-dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HIV infection with HIV RNA < 50 cps/ml within a period of at least 24 weeks suppressive ART prior to randomization, with one accepted blip of HIV RNA < 200 cps/ml and well-tolerated antiretroviral therapy: consisting of 2 NRTI (ABC/3TC, F/TDF or F/TAF) in combination with DRV/r for a period of at least 28 days prior to randomizsation.
* No known genotypic DRV- or integrase inhibitor-related HIV resistance
* Signed written informed consent
* Documented negative HLA B*57:01 (only in case of Abacavir-containing ART)
* A female subject may be eligible to enter and participate in the study if she:

  * is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or
  * is of child-bearing potential with a negative pregnancy test at both screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:
* Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IMP, throughout the study, and for at least 2 weeks after discontinuation of all study medications
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
* Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject
* Approved hormonal contraception without DRV/r interactions and a barrier method
* Any other method with published data showing that the expected failure rate is <1% per year. Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of IMP.

Exclusion Criteria:

* Pregnant women and nursing mothers
* Chronic HBV infection (HBsAg positive); known anti-HBsAb > 10 IU/ml within the last 36 months or a history of infection with known anti-HBcAb positive AND anti-HBsAb > 10 IU/ml AND HBsAg-loss are not exclusionary)
* Any evidence of a Center for Disease Control and Prevention (CDC) Category C disease at screening, except cutaneous Kaposi's sarcoma not requiring systemic therapy. Historical or current CD4 cell counts < 200 cells/mm3 or historic CDC C diseases are not exclusionary
* History or presence of allergy to the study drugs or their components
* Subject has creatinine clearance of <50 mL/min by MDRD eGFR calculation
* Alanine aminotransferase (ALT) ≥ 5 times the upper limit of normal (ULN), OR ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin)
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects with severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification
* Anticipated need for interferon-based Hepatitis C virus (HCV) therapy during the study
* Participation in other interventional clinical trials at the same time
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Persons held in an institution by legal or official order
* Imprisoned people, people requiring in-house treatment for psychiatric disorders or people who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
number (%) of patients with fully suppressed HIV RNA < 50 cps/ml at week 48 | 48 weeks
  For primary endpoint, HIV RNA suppression < 50 cps/ml will be assessed at week 48, using NAT diagnostic.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Spinner, MD, Study Chair — Dep. of Medicine II & IZAR, Klinikum rechts der Isar der TUM
Locations (1):
- Klinikum rechts der Isar, Munich, Germany